CLINICAL TRIAL: NCT07031531
Title: Effectiveness of an AI-Enabled Stratified Management System for Premature Coronary Artery Disease (SMART-CHD): A Prospective, Multicenter, Open-Label, Randomized Controlled Trial
Brief Title: Effectiveness of an AI-Enabled Stratified Management System for Premature Coronary Artery Disease
Acronym: SMART-CHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023ZD0504005
Record Dates: First submitted 2025-05-18; First posted 2025-06-22 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-06

CONDITIONS: Premature Coronary Heart Disease
Keywords: Premature coronary heart disease; secondary prevention; long-term management; mobile health; artificial intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-Enabled Stratified Management Group (Experimental): Participants in the intervention group will use SMART-CHD alongside usual post-discharge care.
  Interventions: Combination Product: AI-Enabled Stratified Management System; Combination Product: Usual Post-Discharge Care
- Usual Post-Discharge Care Group (Active Comparator): Participants in the control group will receive usual discharge protocol comprising verbal and printed discharge instructions addressing medication schedules, follow-up timelines, and lifestyle optimization strategies.
  Interventions: Combination Product: Usual Post-Discharge Care

INTERVENTIONS:
Combination Product: AI-Enabled Stratified Management System — After discharge, participants install SMART-CHD, sync their EHR data, and complete a 10-minute orientation. They then use the app's OCR-assisted surveys to report lifestyle, lab, and event data, while paired wearables stream continuous vitals. AI voice calls and a CRC-managed WeChat group deliver reminders and support. The app's embedded predictive models stratify them into risk tiers and generate tier-specific follow-up schedules. Personalized lifestyle modification guidance, dietary plans, and medication adjustment recommendations are generated by the platform's module. Automated alerts and teleconsultation options are triggered upon detection of high-risk signs or abnormal results, ensuring timely clinical intervention and enhanced secondary prevention.
  Arms: AI-Enabled Stratified Management Group
Combination Product: Usual Post-Discharge Care — Usual discharge protocol comprising verbal and printed discharge instructions addressing medication schedules, follow-up timelines, and lifestyle optimization strategies.

SUMMARY:
The goal of this clinical trial is to learn if an AI-enabled stratified management system (SMART-CHD) can improve post-discharge outcomes in adults aged 18-45 with premature coronary artery disease. The main questions it aims to answer are:

1. Does SMART-CHD reduce the combined rate of all-cause death, myocardial infarction, stroke and rehospitalization within 12 months?
2. Does SMART-CHD achieve better control of modifiable risk factors compared with usual care?

Researchers will compare SMART-CHD to standard discharge management (verbal and printed instructions on medications, follow-up timelines and lifestyle advice) to see if the AI-driven platform leads to fewer adverse events and improved risk-factor profiles.

Participants will:

1. Install and use the SMART-CHD mobile app after a 10-minute structured orientation session with supervised simulations.
2. Complete regular in-app surveys on lifestyle behaviors, laboratory/imaging results and clinical events (with OCR-powered LLM assistance).
3. Wear paired sensors for continuous monitoring of blood pressure, heart rate and other physiologic metrics.
4. Receive automated EHR data harvesting, AI-driven voice-call reminders, and real-time CRC support via a dedicated WeChat group.
5. Follow personalized, guideline-based risk-factor recommendations (diet, exercise, sleep, weight, smoking, alcohol, hypertension, dyslipidemia, diabetes).

ELIGIBILITY:
Inclusion Criteria

1. Patients with coronary heart disease aged 18-45 years;
2. The patient or a close family member is capable of using a smartphone and mobile application (App);
3. Willing to participate in the study and able to provide written informed consent.

Exclusion Criteria

1. Severe cognitive impairment;
2. Advanced-stage malignancy;
3. Life expectancy less than 12 months;
4. Severe multi-organ failure;
5. Refusal to provide written informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4900 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Composite Endpoint Events | Assessed at 12 months post-discharge
  A composite of all-cause death, myocardial infarction, stroke, and unplanned cardiovascular-related rehospitalization.

SECONDARY OUTCOMES:
Individual components of cardiac events | Assessed at 12 months post-discharge
  All-cause death, myocardial infarction, stroke, and unplanned cardiovascular-related rehospitalization
LDL-C level | Assessed at 12 months post-discharge
  Low-density lipoprotein cholesterol level. Unit of Measure: mmol/L.
LDL-C Goal Attainment | Assessed at 12 months post-discharge
  Achieving LDL-C < 1.8 mmol/L.
Blood pressure level | Assessed at 12 months post-discharge
  Systolic blood pressure and Diastolic blood pressure. Unit of Measure: mmHg.
Blood pressure goal attainment | Assessed at 12 months post-discharge
  Achieving target BP <130/80 mmHg.
Hemoglobin A1c level | Assessed at 12 months post-discharge
  Glycated hemoglobin (HbA1c). Unit of Measure: Percentage (%).
Smoking | Assessed at 12 months post-discharge
  Self-reported current smoking status. Unit of Measure: Number and percentage of current smokers
Medication adherence to antiplatelet agents and statins | Assessed at 12 months post-discharge
  Adherence is defined as self-reported use of the medication for more than 80% of the time during the past month

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Fuwai Hospital, Chinese Academy of Medical Sciences/National Center for Cardiovascular Diseases, Beijing, Beijing Municipality
  - Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen, Guangdong
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital Of Hebe Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - Zhengzhou University Affiliated Zhengzhou Central Hospital, Zhengzhou, Henan
  - Zhengzhou University Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shanxi Cardiovascular Disease Hospital, Taiyuan, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in publications will be shared, including all collected de-identified IPD.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 6 months after publication of the primary results and will remain available for at least 5 years thereafter.
Access Criteria: De-identified IPD and supporting documents will be made available upon reasonable request to the Principal Investigator (PI). Requests must include a methodologically sound proposal and intended use. Access will be granted at the discretion of the PI after review of the request.